CLINICAL TRIAL: NCT02444884
Title: A Phase I/II Study of MLN8237, an Oral Selective Small Molecule Inhibitor of Aurora A Kinase, in Children With Relapsed/Refractory Solid Tumors
Brief Title: MLN8237 to Treat Children With Relapsed/Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADVL0812
Record Dates: First submitted 2015-05-07; First posted 2015-05-15 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Unspecified Childhood Solid Tumor, Excluding CNS; Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stratum A1 (Experimental): Establish MTD in patients with solid tumors MLN8237 orally, once daily on Days 1-7
  Interventions: Drug: MLN8237
- Stratum A2 (Experimental): MTD determined in Stratum A1in patients with solid tumors MLN8237 orally, twice daily on Days 1-7
  Interventions: Drug: MLN8237
- Stratum B (Experimental): Expand MTD in patients with neuroblastoma MLN8237 orally, once daily on Days 1-7
  Interventions: Drug: MLN8237

INTERVENTIONS:
Drug: MLN8237
  Other Names: Alisertib

SUMMARY:
RATIONALE: MLN8237 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I/II trial is studying the side effects and best dose of MLN8237 and to see how well it works in treating young patients with relapsed or refractory solid tumors

DETAILED DESCRIPTION:
1.1 Primary Aims 1.1.1 To estimate the maximum tolerated dose (MTD) and recommended Phase II dose of MLN8237 administered orally once daily for 7 days every 21 days to children with refractory solid tumors. 1.1.2 To estimate the maximum tolerated dose (MTD) and recommended Phase II dose of MLN8237 administered orally twice daily for 7 days every 21 days to children with refractory solid tumors. 1.1.3 To define and describe the toxicities of MLN8237 administered on this schedule.

1.1.4 To characterize the pharmacokinetics of MLN8237 in children with refractory cancer.

1.2 Secondary Aims 1.2.1 To preliminarily define the antitumor activity of MLN8237 within the confines of a Phase I study. 1.2.2 To obtain initial Phase II efficacy data on the anti-tumor activity of MLN8237 in children with relapsed-refractory neuroblastoma using the once daily dosing schedule. 1.2.3 To explore the relationship between polymorphic variations in the UDPglucuronyltransferase gene UGT1A1 and exposure to MLN8237.

1.2.4 To assess two common polymorphic variants in the Aurora A kinase gene (Phe31Ile and Val57Ile) thought to potentially influence tumorigenesis. 1.2.5 To preliminarily examine the relationsh

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Patients must have had histologic verification of malignancy at original diagnosis or relapse except in patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevations of CSF or serum tumor markers including alpha-fetaprotein or beta-HCG.
* Performance Level: Karnofsky >/= 50% for patients > 16 years of age and Lansky

  >/= 50 for patients </=16 years of age
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study
* Adequate Bone Marrow Function Defined as:

  a. For patients with solid tumors:
* Peripheral absolute neutrophil count (ANC) >/= 1000/microLiter
* Platelet count >/= 100,000/microLiter (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
* Hemoglobin >/= 8.0 g/dL (may receive RBC transfusions)
* Creatinine clearance or radioisotope GFR >/= 70ml/min/1.73 m2
* Bilirubin (sum of conjugated + unconjugated) </= 1.5 x upper limit of normal (ULN) for age, and
* SGPT (ALT) </= 5.0 x ULN for age (≤ 225 U/L). For the purpose of this study, the ULN for SGPT is 45 U/L.
* Serum albumin >/= 2 g/dL.

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study
* Growth factors that support platelet or white cell number or function must not have been administered within the 7 days prior to enrollment.
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the prior 7 days are not eligible.
* Patients who are currently receiving another investigational drug are not eligible.
* Patients who are currently receiving other anticancer agents, digoxin, cyclosporine, tacrolimus or sirolimus, use of daily benzodiazepines are not eligible
* Patients who have an uncontrolled infection are not eligible.

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose and RP2D administered once daily on Days 1-7 | Up to 21 days (1st cycle) of protocol therapy
Determine maximum tolerated dose and RP2D administered po BID on Days 1-7 | Up to 21 days (1st cycle) of protocol therapy
Adverse events as assessed by (CTCAE) version 4.0 | Every 21 days (each cycle) of protocol therapy for up to 35 cycles [up to 105 weeks]
  DLT will be defined as possibly, probably or definitely attributable to MLN8237. The DLT observation period for the purposes of dose-escalation will be the first cycle of therapy
PK Profile: MLN8237 concentrations in plasma samples | 30 min after the first dose, and at 1,2, 3, 4, 6-8, 24 hours, Day 4 and 7 in Cycle 1
  single-dose AUC, trough estimation, t½ of accumulation

REFERENCES:
- [Derived] Zhou X, Mould DR, Yuan Y, Fox E, Greengard E, Faller DV, Venkatakrishnan K. Population Pharmacokinetics and Exposure-Safety Relationships of Alisertib in Children and Adolescents With Advanced Malignancies. J Clin Pharmacol. 2022 Feb;62(2):206-219. doi: 10.1002/jcph.1958. Epub 2022 Jan 15. PMID 34435684